CLINICAL TRIAL: NCT01709461
Title: Continue Providing Care for Patient Who Participated in the Adagio TVP 1012/501 Clinical Trial
Brief Title: Continuation Treatment Protocol for Patients Who Participated in the Adagio TVP 1012/501 Clinical Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RD 06 - 12
Record Dates: First submitted 2012-10-14; First posted 2012-10-18 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
the purpose of the study is to extend the use of Rasagelin Mesylate 1mg per day by subjects who participated in the Adagio TVP 1012/501 according to form 4a for additional three years.

ELIGIBILITY:
Inclusion Criteria:

* subjects who are willing to contiue this treatment.
* subjects who took part in the TVP 1012/501 clinical trail.

Exclusion Criteria:

* subjects who didn't take part in the TVP 1012/501 clinical trail.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects who took part in the TVP 1012/501 clinical trial and willing to contiue receiving Rasgiline Mesylate.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2012-10

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center Beilinson Campus, Petach Tiqva, Central District, Israel